CLINICAL TRIAL: NCT06200116
Title: Evaluation of a Novel Auto Segmentation Algorithm for Normal Structure Delineation in Radiation Treatment Planning
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ROR2272; NCI-2023-10652 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ROR2272 (Other: Mayo Clinic in Rochester); 22-004438 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Malignant Solid Neoplasm; Hematopoietic and Lymphatic System Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants complete surveys about the performance/functionality of the auto-segmentation algorithm on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study measures the utility of a novel artificial intelligence (AI) algorithm for performing auto-segmentation of computed tomography (CT) scans for radiation therapy planning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To measure the observed utility of an AI algorithm for normal segmentation by recording study subjects' observations of its function.

OUTLINE: This is an observational study.

Participants complete surveys about the performance/functionality of the auto-segmentation algorithm on study.

ELIGIBILITY:
Inclusion Criteria:

* Employment at Mayo Clinic Arizona, Florida, or Rochester (which includes Regional Practice sites located at Mayo Clinic Health System locations) as train clinical staff that participate in normal tissue segmentation

Exclusion Criteria:

* Inability to complete study surveys

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All employed medical dosimetrists or medical dosimetry assistants who routinely perform review of AI generated auto-segmentation of normal tissues.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of success | Baseline
  Will be evaluated by question 1 of the end user survey, which evaluates the level of modification to the artificial intelligence generated auto-segmentation structures that was required (no modification, minor modification, or major modification). Auto-segmentation algorithm data will be collected through an electronic data collection form.

CONTACTS AND LOCATIONS:
Overall Officials: Doug J. Moseley, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials